CLINICAL TRIAL: NCT06311799
Title: Advancing Health Equity by Integrating Social-Clinical Models During Pregnancy
Acronym: FIMPreg
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Geisinger Clinic (Other)
Collaborators: Family Health Council of Central Pennsylvania (FHCCP) (Unknown); American Heart Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2024-0102
Record Dates: First submitted 2024-03-08; First posted 2024-03-15 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Cardiovascular Diseases; Obesity, Maternal; Diabetes
MeSH Terms: conditions — Cardiovascular Diseases; Pregnancy in Obesity; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm 1: Clinic Model (No Intervention): Clinical team gives WIC information only
- Arm 2: Clinic-WIC Model (Active Comparator): Clinical team connects patient to WIC
  Interventions: Behavioral: WIC Referral
- Arm 3: Clinic-RDN Model (Active Comparator): Clinical team gives WIC information only; connects patient to registered dietitian/nutritionist (RDN)
  Interventions: Behavioral: RDN Referral
- Arm 4: Clinic-WIC-RDN (Active Comparator): Clinical team connects patient to WIC and RDN
  Interventions: Behavioral: WIC Referral; Behavioral: RDN Referral

INTERVENTIONS:
Behavioral: WIC Referral — Clinical team will refer study participants to WIC
  Arms: Arm 2: Clinic-WIC Model; Arm 4: Clinic-WIC-RDN
Behavioral: RDN Referral — Clinical team will refer study participants to a RDN
  Arms: Arm 3: Clinic-RDN Model; Arm 4: Clinic-WIC-RDN

SUMMARY:
This study is being done to find out if online referrals to a food management program for Women, Infants, and Children (WIC) made by clinical teams will get more people to enroll in WIC. Women aged 18 or older who get healthcare at Geisinger, are pregnant, and are eligible to be referred to the WIC program will be recruited. These women need to consent to join this study. There are four groups in this study. Group 1 will get usual care with details about WIC from their clinical team. Group 2 will be sent to WIC by their clinical team. The study team may help the clinical team with the referrals. Group 3 will get details about WIC from their clinical team and a dietitian will talk to them about heart-healthy diets and food management. Group 4 will be sent to WIC by their clinical team or study team and a dietitian will talk to them about heart-healthy diets and food management. Participants who talk with the dietitians will be sent kitchen utensils based on need. This study will last about 18 months and will have 240 total subjects joining at about 60 per month. Each subject will be in the study for about 6 months. Subjects will be asked to complete surveys at the start and end of the study. Some subjects will also be asked about their experience in the study after they are done.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Confirmed pregnancy
* Public Insurance (Medicaid) OR no insurance
* If no insurance, must meet income eligibility for WIC
* Intent to deliver at a Geisinger facility
* Able and willing to provide consent

Exclusion Criteria:

* Pre-existing WIC enrollment as a pregnant person
* Not eligible for WIC
* Private insurance
* Unwilling to participate for up to 12 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2024-04-29 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Difference in Women, Infants, and Children (WIC) enrollment | 6 months
  Difference in WIC enrollment between Arm 1 and Arm 3 (Information only) vs Arm 2 and Arm 4 (digital connections)

SECONDARY OUTCOMES:
WIC retention | 6 months
  Number of WIC benefit pick up visits completed
WIC adherence | 6 months
  Frequency of redeeming WIC benefit
Prenatal clinic visit adherence. | 6 months
  Number of prenatal clinic visits attended
Registered Dietitian/Nutritionist (RDN) visit adherence | 6 months
  Number of RDN visits completed

CONTACTS AND LOCATIONS:
Overall Officials: Lisa D Bailey-Davis, Principal Investigator — Geisinger Clinic
Locations (1):
- Geisinger Health System, Danville, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data collected during the trial will be shared, after de-identification.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be made available immediately following publication. No end date.
Access Criteria: Anyone who wishes to access the data may access for any purpose.

REFERENCES:
- [Derived] Herb Neff KM, Brandt K, Chang AR, Lutcher S, Mackeen AD, Marshall KA, Naylor A, Seiler CJ, Wood GC, Wright L, Bailey-Davis L. Comparing models that integrate obstetric care and WIC on improved program enrollment during pregnancy: a protocol for a randomized controlled trial. BMC Public Health. 2024 Dec 5;24(1):3393. doi: 10.1186/s12889-024-20509-6. PMID 39639285